CLINICAL TRIAL: NCT03967600
Title: Clinical and Biological Characteristics of Hidradenitis Suppurativa
Status: Recruiting | Type: Observational
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Other Study IDs: 16-19770
Record Dates: First submitted 2019-05-27; First posted 2019-05-30 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Hidradenitis Suppurativa
MeSH Terms: conditions — Hidradenitis Suppurativa

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Hidradenitis Suppurativa Patients: Patients with physician diagnosed Hidradenitis Suppurativa
- Healthy Volunteers: Healthy volunteers without any skin conditions or recent history of antibiotic use.

SUMMARY:
Hidradenitis suppurativa (HS) is a common and debilitating skin disease that is poorly understood and understudied. As a result, little is known about disease prognosis and few effective treatments exist for this condition. This prospective observational cohort study aims to comprehensively characterize the clinical and biological features of HS. The results of this research will provide a basis for the development of an HS clinical classification system and identification of potential treatments for HS.

ELIGIBILITY:
Hidradenitis Suppurativa Patients

Inclusion Criteria:

1. Age 13 years or older
2. Diagnosis of HS clinically-confirmed by a physician

Exclusion Criteria:

1. Inability to give informed consent or have a parent/guardian who is able and willing to give informed consent.

Healthy Volunteer

Inclusion Criteria:

1. No history of chronic skin conditions
2. No recent history of antibiotic use

Exclusion Criteria:

1. Inability to give informed consent or have a parent/guardian who is able and willing to give informed consent.

Min Age: 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients with Hidradenitis Suppurativa
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2016-07-15 (Actual); Primary Completion 2026-07-15 (Estimated); Study Completion 2026-07-15 (Estimated)

PRIMARY OUTCOMES:
The primary aim of this study is to identify clinical and biologic characteristics of hidradenitis suppurativa. | 2016-2026

SECONDARY OUTCOMES:
Secondary aims include correlating alterations in clinical and biological characteristics with disease status, and identifying genetic variants that predict disease progression or response to therapy. | 2016-2026

CONTACTS AND LOCATIONS:
Overall Officials: Haley B Naik, MD, MHSc, FAAD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No